CLINICAL TRIAL: NCT07398326
Title: Phase II Study of Anlotinib Combined With Sintilimab as First-line Treatment for Advanced Non-liver Metastatic Colorectal Cancer
Brief Title: Anlotinib Combined With Sintilimab as First-line Treatment for Advanced Non-liver Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhan Wang, Department of medical oncology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APICAL-CRC2
Record Dates: First submitted 2026-01-13; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: anlotinib and sintilimab

INTERVENTIONS:
Drug: anlotinib and sintilimab — anlotinib combined with sintilimab as first-line treatment for advanced non-liver metastatic colorectal cancer

SUMMARY:
Colorectal cancer (CRC) is the third most common malignant tumor worldwide and the second leading cause of cancer-related deaths. Despite recent progress in CRC research, approximately 15% to 30% of patients have metastatic lesions at the time of initial diagnosis, and another 20% to 50% of patients with primary localized CRC eventually develop metastatic disease. The conventional treatment for first-line metastatic colorectal cancer (mCRC) is chemotherapy based on fluorouracil combined with anti-EGFR/VEGF targeted drugs. However, some mCRC patients may not be able to receive standard dual or triple chemotherapy combined with targeted therapy due to factors such as advanced age, poor physical condition, comorbidities, or personal preferences. Therefore, exploring new, highly effective, and low-toxicity treatment regimens is of significant clinical importance. The combination of immune checkpoint inhibitors and antiangiogenic TKIs is expected to form a strong synergistic antitumor effect, which opens up a new approach for "chemotherapy-free" treatment of mCRC when the immune system is functioning normally. Previously, we conducted the APICAL-CRC study, enrolling a total of 30 patients. The clinical objective response rate (ORR) was 48.3%, the disease control rate was 89.7%, and the median progression-free survival (mPFS) and median overall survival (mOS) were 8.6 months and 22.9 months, respectively. Subgroup analysis later revealed that the ORR for non-liver metastasis patients was 70%, with an mPFS of 14.9 months, significantly higher than that of liver metastasis patients (ORR 36.8%). At the same time, patients with better physical performance scores (ECOG PS 0-1) had an ORR of 66.7%, which was superior to that of patients with ECOG PS 2 (21.4%). In terms of safety, the incidence of grade ≥ 3 treatment-related adverse events (TRAEs) for the combination of anlotinib and sintilimab was only 13.3%. Based on the preliminary results of the APICAL-CRC study, we consider further precise screening of the advantageous population among advanced CRC patients for subsequent research. We plan to limit the enrolled patients to those without liver metastasis and with ECOG PS 0-1, providing new strategies and methods for precise treatment of advanced CRC.The purpose of this study is to evaluate the efficacy and safety of anlotinib combined with sintilimab as first-line treatment for non-liver metastatic advanced colorectal cancer. The study will be conducted at Shanghai Changzheng Hospital. The study drugs, anlotinib and sintilimab, are both marketed drugs in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced colorectal adenocarcinoma.
* Patients with non-hepatic metastases who explicitly refuse chemotherapy.
* Patients who have not received prior systemic therapy, or those with metastasis or recurrence occurring ≥12 months after completion of adjuvant therapy.
* At least one measurable lesion according to RECIST 1.1 criteria.
* Prior local radiotherapy is permitted if completed at least 3 weeks before the first study drug administration; however, lesions used for RECIST evaluation must be outside the radiation field.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Ability to understand and voluntarily provide written informed consent.
* For women of childbearing potential, a negative pregnancy test within 7 days prior to treatment initiation. Both patients and their partners must agree to use effective contraception during the study period.

Exclusion Criteria:

* Patients who have undergone major surgery or sustained severe trauma within 4 weeks prior to the first dose of the study drug.
* Patients with a history of hypersensitivity to any component of the study regimen.
* Patients who are planning to conceive, are pregnant.
* Patients with brain metastases who are unable to accurately describe their symptoms or condition.
* Patients with a history of autoimmune diseases or organ transplantation.
* Use of immunosuppressive medications within 2 weeks prior to the initiation of study treatment (excluding inhaled corticosteroids, or physiological replacement doses of steroids equivalent to ≤10 mg/day of prednisone).
* Administration of a live attenuated vaccine within 4 weeks prior to the start of study treatment or planned vaccination during the study period.
* Prior treatment with anlotinib, anti-PD-1/PD-L1 monoclonal antibodies, or any other therapy targeting T-cell co-stimulation or immune checkpoint pathways.
* History of any of the following within 6 months before starting study treatment: myocardial infarction, severe/unstable angina, congestive heart failure of New York Heart Association (NYHA) Class 2 or higher, or poorly controlled cardiac arrhythmias.
* Laboratory test abnormalities meeting any of the following criteria:

  1. Absolute neutrophil count (ANC) <1,500/mm³.
  2. Platelet count <75,000/mm³.
  3. Total bilirubin >1.5 times the upper limit of normal (ULN).
  4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 times ULN.
  5. Serum creatinine >1.5 times ULN.
* Diagnosis of any malignancy other than advanced colorectal cancer within the 5 years preceding the start of study treatment, except for carcinoma in situ of the cervix, cured basal cell carcinoma, or bladder epithelial tumors.
* Patients with colorectal cancer amenable to curative surgical resection (however, those who explicitly refuse surgery or are deemed unsuitable for surgery may be eligible).
* History of substance abuse, drug use, or alcohol dependence.
* Lack of legal capacity or limited civil capacity.
* Any other condition that, in the opinion of the Investigator, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Naval Medical University, Shanghai, China

DOCUMENTS (2):
  • Study Protocol (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT07398326/Prot_000.pdf
  • Informed Consent Form (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT07398326/ICF_001.pdf